CLINICAL TRIAL: NCT06913959
Title: HIV-1 Non-group M in Cameroon : Study of Genotypic and Phylogenetic Diversity (OBSOCAM)
Acronym: OBSOCAM
Status: Not yet recruiting | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University Hospital, Rouen (Other); Centre Pasteur du Cameroun (Other)
Responsible Party: Sponsor
Other Study IDs: ANRS0098s
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: HIV Infection
Keywords: HIV genetic diversity; HIV-1 non-M variants
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples, 2x 5ml EDTA (ethylenediaminetetraacetic acid)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Dried Blood Spot samples tested positive for HIV during the previous national epidemiologic surveys Demographic health surveys in Cameroon
  Interventions: Diagnostic Test: Prospective
- Prospective: Individuals who came to Center Pasteur in Yaounde or Garoua for HIV screening or viral load monitoring
  Interventions: Diagnostic Test: Prospective

INTERVENTIONS:
Diagnostic Test: Prospective — Blood samples will be collected in order to meet the objectives of this substudy and possibly for complementary research

SUMMARY:
The aim of the study is to study the genotypic characteristics of HIV-1 non-M circulating in the whole Cameroon and their genetic evolution.

DETAILED DESCRIPTION:
HIV-1 is divided four distinct groups: M (major) which represents the pandemic strains while others groups O (outlier), N (non M, non O) and P are called non-M variants. Group O (HIV-O) is more divergent, endemic in Central Africa and Cameroon, where it represents about 1% of HIV infections. These variants are characterized by an important genetic divergence from pandemic HIV-1 group M (HIV-M), which impacts on the diagnosis, monitoring and treatment of infected patients. Although discovered in 1990, and emerged at the same time as HIV-M, no data of epidemiology, natural history and evolution of the genetic diversity of these variants is currently available. The few knowledge available to date come from sporadic cases, mainly through studies in Yaoundé. It is therefore essential to improve current knowledge on these variants and their consequences on infected patients.

The aim of the study is to study the genotypic characteristics of HIV-1 non-M circulating in the whole Cameroon and their genetic evolution.

ELIGIBILITY:
Inclusion Criteria:

* All available samples tested positive for HIV during the national Health survey of Cameroon in 2011 And 2018
* All Individuals who came to Centre Pasteur in Yaoundé or Garoua for HIV screening or viral load monitoring.

Exclusion Criteria:

* Insufficient quantity or degraded Dried Blood Spot samples
* All HIV-positive individuals aged less than 21 years, infected with a Group M HIV-1 virus, or those who refused to participate in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective phase : Dried Blood Spot samples tested positive for HIV during the Demographic health surveys in Cameroon 2011 and 2018 surveys, serotyping for HIV.
  Prospective phase : Individuals who came to Center Pasteur Cameroon in Yaoundé or Garoua for HIV screening or viral load monitoring, serotyping of HIV for positive samples.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of non-M HIV-1 in Cameroon | 1 day
  Number of participants infected with non-M HIV-1 included compared to the total expected number of inclusions

SECONDARY OUTCOMES:
Investigate the current molecular epidemiology of resistance in non-M HIV-1 variants in Cameroon | 1 Day
  Proportion of non-M HIV-1 samples characterized genotypically among the samples collected from participants included in the project

OTHER OUTCOMES:
Study the current molecular epidemiology of HIV 1 non-M variant resistance in Cameroon | 1 day
  Proportion of non-M HIV-1 samples characterized for resistance among the samples collected from participants included in the project

IPD SHARING:
Plan to Share IPD: No